CLINICAL TRIAL: NCT06248333
Title: Subthalamic Nucleus Electrical Stimulation for Drug-resistant Focal Motor Epilepsy: A Multicenter, Randomized, Double-blind, Sham-controlled, Parallel-group Trial
Brief Title: Subthalamic Nucleus Electrical Stimulation for Drug-resistant Focal Motor Epilepsy
Acronym: STEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Sanbo Brain Hospital (Other); Qilu Hospital of Shandong University (Other); Peking University (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-174-002
Record Dates: First submitted 2024-01-14; First posted 2024-02-08 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy, Drug Resistant
Keywords: Deep Brain Stimulation; Drug Resistant Epilepsy; Subthalamic Nucleus; Focal Motor Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy, Partial, Motor

STUDY DESIGN:
Intervention Model Description: After completion of DBS surgery (Month 0), participants will undergo an 8-day parameter exploration period after 1-month postoperative recovery (month 1), and DBS off after individual parameters have been determined. At Month 2, participants will be randomly assigned to one of two groups: Group A or Group B. Group A (Activate Stimulation) will have their stimulator turned on after randomization. Group B (Sham Stimulation) will receive sham stimulation, meaning the stimulator will remain off until Study Month 5. At Month 5, Group A will continue to receive stimulation and not have the stimulator turned off, and the stimulator in Group B will be turned on and left on for the remainder of the study (Month 11).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One day before the first programming, the grouper and the programmer will release the cover independently. Only the grouper and the programmer will know the group information of each patient, in which the programmer does not communicate with the patient about the programming parameters. After each programming, the results are uniformly placed in the programmer to keep the others (patients, neurologists) blind about grouping and parameters. The evaluation will be finished by neurologists, who do not participate in the surgical treatment and programmer. So that the participants, care providers, investigators, and outcomes assessors will not know which group are assigned to from randomization (Month 2) to Month 5. The statistical team is independent of other researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Stimulation (Experimental): After randomization, participants will undergo STN-DBS ON in the 3-month blinded phase (Month 2 to Month 5) with the individual stimulation parameters determined in the parameter determination period, then continue to receive stimulation for the remainder of the study.
  Interventions: Device: STN-DBS ON
- Sham Stimulation (Sham Comparator): After randomization, participants will undergo STN-DBS OFF in the 3-month blinded phase (Month 2 to Month 5) with 0mA current, then the stimulator will be turned on with individual stimulation parameters and left on for the remainder of the study.
  Interventions: Device: STN-DBS OFF

INTERVENTIONS:
Device: STN-DBS ON — Stimulation ON
  Arms: Active Stimulation
Device: STN-DBS OFF — Stimulation OFF
  Arms: Sham Stimulation

SUMMARY:
The primary objective of this research is to study the efficacy and safety of deep brain stimulation (DBS) of subthalamic nucleus (STN) as adjunctive therapy for reducing the frequency of seizures in drug-resistant focal motor epilepsy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, sham-controlled, parallel-group trial that aims to investigate the efficacy of STN-DBS in reducing the frequency of seizures in drug-resistant focal motor epilepsy. Participants who were eligible for the inclusion criteria and ineligible for the exclusion criteria will be randomly assigned into two groups by a 1:1 ratio. The primary purpose of this study is to compare active STN-DBS with sham STN-DBS in reducing seizure frequency. Both intent analysis (ITT) and compliance program set (PPS) were used for analysis. Only high-volume centers with a proven track record will be included. The STEM trial will be conducted in 5 sites in China.

ELIGIBILITY:
Inclusion Criteria:

* 14-65 years of age, inclusive, at Screening Visit.
* Refractory to anti-seizure medications (ASMs).
* Diagnosed with focal motor epilepsy, which meets the following items:

  1. Seizure mainly presents as focal tonic, myoclonic, or primary motor seizure (including primary sensory seizure), with or without secondary bilateral tonic-clonic seizure.
  2. After a comprehensive evaluation, the epileptogenic zone was presumed to predominantly involve the unilateral or bilateral central area (precentral gyrus, postcentral gyrus, and paracentral lobule) or supplementary motor area according to comprehensive presurgical evaluation.
* Within 1 month prior to the Screening Visit (M-3), the following conditions are met:

  1. At least 3 focal onset seizures (with or without secondary bilateral tonic-clonic seizure).
  2. Subject is receiving at least one type of ASM[s], and the regimen has been stable (no addition or removal of ASM[s] [not counting brief rescue medicines such as benzodiazepines]; dose adjustments are permitted to ASM[s]).
* Within the baseline period (3 months after the Screening Visit [M-3]), the following conditions are met:

  1. The patient or their caregiver is capable of completing the seizure diary.
  2. Seizure diary shows an average of 3 or more partial-onset seizures (with or without secondary bilateral tonic-clonic seizure) per month during the Baseline Period, with no more than 30 days between seizures.
  3. The regimen of ASM[s] has been stable (no addition or removal of ASM[s] [not counting brief rescue medicines such as benzodiazepines]; dose adjustments are permitted to ASM[s]).
* After comprehensive preoperative evaluation, patients who are considered unsuitable for or refuse resection surgery, or those for whom the effects of epileptic focus resection and thermocoagulation surgery are not satisfactory.
* Informed consent signed.

Exclusion Criteria:

* Diagnosed with generalized or hereditary epilepsy with ion channel gene mutations;
* Seizures mainly present as complex motor seizures (e.g., hyperkinetic, automatisms, etc.);
* Tonic-clonic status epilepticus within12 months;
* Psychogenic non-epileptic seizures within 12 months;
* Structural lesion of the subthalamic nucleus;
* Presence of implanted electrical stimulation medical device anywhere in the body (e.g., pacemaker, spinal cord stimulator, responsive neurostimulation) or any metallic implants in the head (e.g., aneurysm clips, cochlear implants). Note: Vagal nerve stimulators are allowed if the parameter remains stable for at least 3 months prior to the screening visit;
* Risk factors that would put the participant at risk for intraoperative or postoperative bleeding. (e.g., coagulation abnormalities, etc.) or the need for chronic anticoagulation or antiplatelet aggregation medications;
* IQ < 55 or severe cognitive dysfunction, unable to complete the study;
* Diagnosed with a progressive neurological disorder (including progressive Rasmussen's encephalitis, etc.);
* Diagnosed with a severe neuropsychiatric disorder such as dementia, major depression (admission to a psychiatric specialty/hospital within 5 years or any suicidal or self-injurious tendencies), schizophrenia, or neurodegenerative disorders;
* Diagnosed with other serious physical disorders, internal diseases or severe abnormalities in liver or kidney function;
* Pregnant, or planning to pregnant within 2 years;
* Participation in another clinical study within 3 months;
* Not suitable for enrollment as assessed by the multidisciplinary team of the center.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Median Percent Change in Seizure Frequency | Through the end of the three-month blinded phase
  Seizure frequency (SF28) is defined as seizure count per month (28-day) period. The SF28 is calculated as follows, where D=total number of days for which seizure information is collected for the specific 28-day interval:
  SF28=(Total number of seizures in D days/D)*28. In addition, the baseline seizure frequency is defined as mean of 3-month SF28 in the baseline period. The seizure frequency in double-blind phase is defined as SF28 per month during the double-blind period. Percent change in seizure frequency=100*(double-blind SF28-baseline SF28)/baseline SF28.

SECONDARY OUTCOMES:
Seizure Responder Rate | Through the end of the three-month blinded phase
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Seizure Severity | Through the end of the three-month blinded phase
  The percent change from baseline in seizure severity evaluated by Liverpool seizure severity scale (LSSS) across the double-blind period.
Seizure-free Days | Through the end of the three-month blinded phase
  Change in percentage of seizure-free days over the entire blinded phase as compared to the entire baseline phase. The number of seizure-free days was normalized to 84-day baseline and blinded phases for each subject.
The maximum length of seizure-free Intervals | Through the end of the three-month blinded phase
  Percentage change in the maximum length of seizure-free intervals over the entire blinded phase as compared to the entire baseline phase.
Life quality evaluation | Through the end of the three-month blinded phase
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score at 3 months after randomization.
Motor function evaluation | Through the end of the three-month blinded phase
  Percentage change from baseline in Unified Parkinson's Disease Rating Scale part II & part III (UPDRS II-III) score at 3 months after randomization.
Cognitive function evaluation (MMSE) | Through the end of the three-month blinded phase
  Percentage change from baseline in Mini-Mental State Examination (MMSE) score at 3 months after randomization.
Cognitive function evaluation (MoCA) | Through the end of the three-month blinded phase
  Percentage change from baseline in Montreal Cognitive Assessment (MoCA) score at 3 months after randomization.
Psychologic Evaluation (Anxiety) | Through the end of the three-month blinded phase
  Percentage change from baseline in Hamilton Anxiety Rating Scale (HAMA) score at 3 months after randomization.
Psychologic Evaluation (Depression) | Through the end of the three-month blinded phase
  Percentage change from baseline in Hamilton Depression Rating Scale (HAMD) score at 3 months after randomization.
Sleep Quality | Through the end of the three-month blinded phase
  Percentage change from baseline in Pittsburgh Sleep Quality Index (PSQI) score at 3 months after randomization.
Adverse Events | Through Month 11 of the open-label follow-up phase
  Rate of adverse events which were judged to be study-related throughout the study.
Incidence of Sudden Unexpected Death in Epilepsy (SUDEP) | Through Month 11 of the open-label follow-up phase
  The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No